CLINICAL TRIAL: NCT07109297
Title: A Phase 4, Open-label, Single-arm Clinical Study to Describe Safety and Efficacy Outcomes Associated With the Use of Nirsevimab in Neonates and Infants Born During or Entering Their First Respiratory Syncytial Virus (RSV) Season and in Children up to 24 Months of Age Who Remain Vulnerable to Severe RSV Disease Through Their Second RSV Season
Brief Title: Study of Monoclonal Antibody Nirsevimab Against Respiratory Syncytial Virus (RSV) in Participants up to 24 Months of Age in India
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VAS00017; U1111-1310-0978 (Other: WHO ICTRP)
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: RSV Immunization
MeSH Terms: interventions — nirsevimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nirsevimab (Experimental): Participants will receive:
  * 1 intramuscular (IM) injection for neonates and infants aged 0 to 12 months born or entering their first RSV season at Day 01
  * 2 IM injections for children up to 24 months of age who remain vulnerable to severe RSV disease through their second RSV season at Day 01
  Interventions: Biological: Nirsevimab

INTERVENTIONS:
Biological: Nirsevimab — Pharmaceutical form:Sterile solution for injection-Route of administration:Intramuscular
  Other Names: 526; Beyfortus®

SUMMARY:
The purpose of this study is to describe the safety and efficacy outcomes associated with the use of nirsevimab, administered as per routine clinical practice, in neonates and infants aged 0 to 12 months born during or entering their first RSV season and in children up to 24 months of age who remain vulnerable to severe RSV disease through their second RSV season.

DETAILED DESCRIPTION:
Study duration: up to 16 months, including 10 months of enrollment and 6 months of follow-up

* Treatment duration: 1 day; 1 intramuscular (IM) injection
* Visit frequency:

  * 1 in-person visit for immunization (Visit [V] 01) at Day (D) 1.
  * 3 phone call visits (V2, V3 and V4) at D31 (+ 14 days), D91 (+ 14 days) and D181 (+14 days) respectively.

ELIGIBILITY:
Inclusion Criteria: - Neonates and infants aged 0 to 12 months on the day of inclusion and born during or entering their first RSV season OR children up to 24 months of age on the day of inclusion who remain vulnerable to severe RSV disease through their second RSV season

Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study intervention used in the study or to a product containing any of the same substances
* Known thrombocytopenia, as reported by the parent(s)/legally acceptable representative(s), contraindicating intramuscular injection
* Known bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular injection
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Active LRTI on the day of study intervention administration
* Active RSV infection on the day of study intervention administration
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of study intervention administration. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Receipt of palivizumab or other RSV monoclonal antibody or any RSV vaccine in the same RSV season than inclusion in the study
* Mother of the participant was administered an RSV vaccine during her pregnancy with the participant
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Receipt of any investigational drug in the last 30 days prior to the inclusion in the study
* Participation at the time of study enrollment or in the 4 weeks preceding the study intervention administration or planned participation during the present study period, in another clinical study investigating a vaccine, drug, medical device, or medical procedure Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Presence of immediate adverse events (AEs) | Within 30 minutes after immunization
  Number of participants experiencing immediate AEs
Presence of non-serious AEs | From Day 01 through Day 31
  Number of participants experiencing non-serious AEs
Presence of adverse events of special interest (AESIs) throughout the study | Throughout the study (approximately 6 months)
  Number of participants experiencing AESIs
Presence of medically attended adverse events (MAAEs) throughout the study | Throughout the study (approximately 6 months)
  Number of participants experiencing MAAEs
Presence of serious adverse events (SAEs) throughout the study | Throughout the study (approximately 6 months)
  Number of participants experiencing SAEs

SECONDARY OUTCOMES:
Incidence of medically attended lower respiratory tract infection (LRTI) (outpatient and inpatient) due to reverse transcription--polymerase chain reaction (RT-PCR) confirmed RSV | Through 180 days after dosing
  Incidence of medically attended LRTI (outpatient and inpatient) due to reverse transcription--polymerase chain reaction (RT-PCR) confirmed RSV
Incidence of LRTI hospitalizations due to RT-PCR confirmed RSV through 180 days after dosing | Through 180 days after dosing
  Incidence of LRTI hospitalizations due to RT-PCR confirmed RSV through 180 days after dosing

CONTACTS AND LOCATIONS:
Locations (7):
- India (7):
  - Investigational Site Number : 3560002, Bengaluru
  - Investigational Site Number : 3560008, Jaipur
  - Investigational Site Number : 3560003, Kolkata
  - Investigational Site Number : 3560007, Nagpur
  - Investigational Site Number : 3560001, New Delhi
  - Investigational Site Number : 3560004, Pune
  - Investigational Site Number : 3560006, Vizianagaram

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VAS00017 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26792&tenant=MT_SNY_9011